CLINICAL TRIAL: NCT03069846
Title: Collecting Spectral Signatures of Melanoma, Squamous Cell Carcinoma, Basal Cell Carcinoma, Benign Lesions and Normal Tissues Using Spectra-Scope
Brief Title: Diagnosing Melanoma, Squamous Cell Carcinoma and Basal Cell Carcinoma Using the Spectra-Scope
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sung Hyun Pyun (Industry)
Responsible Party: Sponsor-Investigator, Sung Hyun Pyun, CEO, Speclipse Australia Pty Ltd
Organization: Speclipse Australia Pty Ltd (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Speclipse-2016-10
Record Dates: First submitted 2017-02-20; First posted 2017-03-03 (Actual); Last update posted 2018-04-20 (Actual); Status verified 2018-04

CONDITIONS: Skin Cancer
Keywords: skin cancer; laser spectroscopy; non-invasive diagnostics
MeSH Terms: conditions — Skin Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Measurement using Spectra-Scope (Experimental): Short pulsed Nd:YAG laser irradiation onto the skin lesion / measurement with Spectra-Scope
  Interventions: Device: Spectra-Scope

INTERVENTIONS:
Device: Spectra-Scope — The Spectra-Scope consists of the light collection module and the spectral analysis module.
  The light collection module is attached to the handpiece of short pulse Nd:YAG laser, and the analysis module is placed on the laser.
  Each potential skin cancer site, which has previously been identified as requiring biopsy, should be assessed using five laser shots that last approximately 10 milliseconds per shot and measurement. The laser shots must be made before the scheduled biopsy.
  All potentially cancerous lesions (or lesions that would usually undergo complete biopsy of the lesion or require follow up within three months) should be sampled. The Spectra-Scope will not provide a diagnosis at the time of sampling. Sites should record the spectra reported for each laser shot in the CRF.

SUMMARY:
The primary objective is to collect emission spectra of normal tissue, pigmented normal lesion, benign lesion, SCC, BCC and melanoma to construct the database and validate the classifying algorithm.

DETAILED DESCRIPTION:
The Speclipse Spectra-Scope consists of the light collection module and the spectral analysis module. The light collection module is attached to the handpiece of short pulse (a few nanoseconds) Nd:YAG (neodymium-doped yttrium aluminium garnet) commercial cosmetic laser, and the analysis module is placed on the laser. When Nd:YAG laser is irradiated onto the skin lesion, the laser ablates a trace amount of tissue, producing micro plasma. The emitted light from the micro plasma is analysed spectrally to determine the elemental and molecular information from the tissue in real time. No calibration of the Spectra-Scope is required.

Before the skin is irradiated with the laser, select the age, sex and the position of the target skin lesion and put the patient number of the day on the software panel of laptop which is connected to the device. Prior to sampling, the skin site must be wiped with ethanol and allowed to air dry. When the laser is irradiated, the emission spectra of tissue is automatically generated from the spectrometer inside the device and simultaneously displayed on the monitor, and stored in the laptop. The spectral data stored in the laptop is wirelessly accessible using Google drive.

An algorithm then determines whether the skin is from a normal, pigmented normal, benign, squamous cell carcinoma (SCC), basal cell carcinoma (BCC) or melanoma based on the spectral 'signature'. These algorithms have been determined during clinical ex-vivo and in-vivo studies performed in Korea. The purpose of this study is to collect tissue emission spectra of Australian patients and to further refine the algorithms, and to confirm the appropriate spectra for 'normal', 'benign', 'melanoma', 'SCC', and 'BCC'.

Each potential skin cancer site, which has previously been identified as requiring biopsy, is assessed using five laser shots that last approximately 10 milliseconds per shot and measurement. The laser shots are made before the scheduled biopsy.

Some of the potential skin cancer sites will be labelled as cancers ('melanoma', 'SCC' or 'BCC') from the biopsy result, and some of the potential skin cancer site will be labelled as 'benign' (control group 1) from the biopsy result.

ELIGIBILITY:
Inclusion Criteria:

1. Be aged 18 years or over;
2. Have at least one suspicious lesion that:

   1. Is required to be biopsied for assessment of skin cancer (as assessed by at least one dermatologist);
   2. Has a diameter of more than 2 mm but less than 22 mm;
   3. Is accessible to the Spectra-Scope device;
3. Provide written informed consent.

Exclusion Criteria:

1. Have a known allergy to ethanol;
2. Have a lesion that:

   1. Has previously been biopsied, excised or traumatised;
   2. Is not intact;
   3. Is within 1 cm of the eye;
   4. Is on a mucosal surface (lips, genitals);
   5. Is on palmar hands;
   6. Is on palmar feet;
   7. Is on or under nails;
   8. Is located on or in an area of visible scarring;
   9. Contains foreign matter (tattoo, splinter, marker)
3. Have an active infection;
4. Have an open lesion sampled;
5. Have an autoimmune disease such as lupus or scleroderma vitiligo.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2017-06-05 (Actual); Primary Completion 2018-06-18 (Estimated); Study Completion 2018-06-18 (Estimated)

PRIMARY OUTCOMES:
The primary endpoint is to compare the aggregated emission spectra of skin cell carcinoma verses normal skin. | We plan to recruit 150 patients within a 3 month time frame.
  The aggregated emission spectra collected over a range of wavelengths from skin cells (skin cancer verses normal skin) irradiated with a commercial laser will be plotted to identify wavelengths with greatest spectra seperation.

CONTACTS AND LOCATIONS:
Overall Officials: Saleem Loghdey, M.D., Principal Investigator — Integrated Specialist Healthcare
Locations (1):
- Integrated Specialist Healthcare, Miranda, New South Wales, Australia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: International Conference of Harmonisation, International Conference on Harmonisation of Technical Requirements for Registration of Pharmaceuticals for Human Use — https://www.ich.org/fileadmin/Public_Web_Site/ICH_Products/Guidelines/Efficacy/E2F/Step4/E2F_Step_4.pdf
- See also: Dickson, P.V. and J.E. Gershenwald, Staging and prognosis of cutaneous melanoma. Surg Oncol Clin N Am, 2011. 20(1): p. 1-17. — https://www.ncbi.nlm.nih.gov/pubmed/21111956
- See also: Rosado, B., Accuracy of Computer Diagnosis of Melanoma. Archives of Dermatology, 2003. 139(3): p. 361. — https://www.ncbi.nlm.nih.gov/pubmed/12622631
- See also: Abbasi, N.R., et al., Early diagnosis of cutaneous melanoma: revisiting the ABCD criteria. JAMA, 2004. 292(22): p. 2771-6. — https://www.ncbi.nlm.nih.gov/pubmed/15585738
- See also: ISO, Clinical investigation of medical devices for human subjects - good clinical practice. ISO 14155:2011 (E). 2011. — http://www.iso.org/iso/catalogue_detail?csnumber=45557